CLINICAL TRIAL: NCT01425554
Title: Doppler Sonography, Magnetic Resonance Venography, Air-plethysmography in the Non-invasive Diagnostics of Chronic Cerebrospinal Venous Insufficiency (CCSVI)
Brief Title: Doppler Sonography, MR Venography, Plethysmography for the Diagnosis of CCSVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Euromedic Specialist Clinics, Poland (Other)
Responsible Party: Principal Investigator, Marian Simka, senior consultant, Euromedic Specialist Clinics, Poland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20/2011
Record Dates: First submitted 2011-08-28; First posted 2011-08-30 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Cerebrospinal Venous Insufficiency
Keywords: Vascular malformations in the internal jugular veins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic study (No Intervention)
  Interventions: Other: Doppler sonography of internal jugular veins; Other: Magnetic resonance venography of internal jugular veins; Other: Air-plethysmography of the neck; Other: Catheter venography of internal jugular veins

INTERVENTIONS:
Other: Doppler sonography of internal jugular veins — Doppler sonography of internal jugular veins
Other: Magnetic resonance venography of internal jugular veins — Magnetic resonance venography of internal jugular veins
Other: Air-plethysmography of the neck — Air-plethysmography of the neck
Other: Catheter venography of internal jugular veins — Catheter venography of internal jugular veins

SUMMARY:
This study is aimed at evaluation of diagnostic value of Doppler sonography, MR venography and air-plethysmography for the assessment of abnormalities in the internal jugular veins, with catheter venography as the reference test.

ELIGIBILITY:
1. Patients group

   Inclusion Criteria:
   * confirmed diagnosis of multiple sclerosis

   Exclusion Criteria:
   * coexisting another neurologic pathology (e.g. stroke, Parkinson disease)
   * significant stenosis of carotid or vertebral arteries
   * other significant abnormalities of blood vessels of the upper part of the body
   * tricuspid valve incompetence
   * allergy to iodine contrast dye
   * chronic renal failure
   * pregnancy
   * other severe comorbidities or significant abnormalities in standard lab tests
2. Healthy volunteers.

Inclusion Criteria:

* none

Exclusion Criteria:

* confirmed diagnosis of multiple sclerosis or related pathologies (CIS, NMO)
* coexisting another neurologic pathology (e.g. stroke, Parkinson disease)
* significant stenosis of carotid or vertebral arteries
* other significant abnormalities of blood vessels of the upper part of the body
* tricuspid valve incompetence

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Positive and negative predictive value of Doppler sonography, MR venography and air-plethysmography | All non-invasive test are done up to 14 days prior to catheter venography
  Positive and negative predictive value of Doppler sonography,MR venography and air-plethysmography for the detecting of vascular malformation in the internal jugular veins with catheter venography as the reference test

CONTACTS AND LOCATIONS:
Locations (1):
- Euromedic Specialis Clinics; ul. Rolna 18, Katowice, Poland